CLINICAL TRIAL: NCT04361292
Title: Effect of Ejaculatory Abstinence Period on Sperm DNA Fragmentation and Pregnancy Outcome of Intrauterine Insemination Cycles: A Prospective Randomized Study
Brief Title: Ejaculatory Abstinence in IUI Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Cihan Kabukcu, Assistant Professor, M.D., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 60116787-020/17327
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Infertility; Spermatozoa; Reproductive Disorder
Keywords: Intrauterine insemination; Ejaculatory abstinence; sperm DNA fragmentation; TUNEL assay
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: One hundred twenty eligible couples were prospectively randomized into two groups on the second day of the cycle just before starting the treatment protocol. Randomization was performed according to a computer-generated random number list at a ratio of 1:1. From the randomization list, an independent secretary who was blind to patients' identities applied the allocation in consecutive order. Patients allocated into group A, had an ejaculatory abstinence period of one day, whereas patients allocated into group B had an ejaculatory abstinence period of three days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: From the randomization list, an independent secretary who was blind to patients' identities applied the allocation in consecutive order. Patients allocated into group A, and group B. Care provider and investigator were blind to patient groups. Participants were informed about the timing of abstinence intervals, but they did not know which groups they were allocated to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: one day abstinence period (Active Comparator): Patients allocated into group A had an ejaculatory abstinence period of one day
  Interventions: Procedure: INTRAUTERINE INSEMINATION
- Group B: three days abstinence period (Active Comparator): Patients allocated into group B had an ejaculatory abstinence period of three days
  Interventions: Procedure: INTRAUTERINE INSEMINATION

INTERVENTIONS:
Procedure: INTRAUTERINE INSEMINATION — Intrauterine insemination (IUI) combined with ovarian stimulation, has been an extensively used procedure for the treatment of patients with unexplained infertility. The fact that IUI is less expensive, less invasive, and easier to perform than other assisted reproductive techniques makes it the first-line treatment option in infertility treatments. Sperm that have been washed and concentrated are placed directly into the uterus around the time of ovulation. All patients had ovulation induction with gonadotropins and ovulation was triggered by recombinant hcg.

SUMMARY:
Intrauterine insemination (IUI) combined with ovarian stimulation, has been an extensively used procedure for the treatment of patients with unexplained infertility. The aim of this study was to report the effect of ejaculatory abstinence on sperm DNA fragmentation and pregnancy rates in IUI cycles, as well as the correlation between the two.

DETAILED DESCRIPTION:
Intrauterine insemination (IUI) combined with ovarian stimulation, has been an extensively used procedure for the treatment of patients with unexplained infertility. The fact that IUI is less expensive, less invasive, and easier to perform than other assisted reproductive techniques makes it the first-line treatment option in infertility treatments. Several studies have been published over the past few years examining the relationship between sperm DNA fragmentation and IUI outcome. The optimal period for ejaculatory abstinence before the semen sample is a controversial issue in the literature. There are only two retrospective studies examining the relationship between the ejaculatory abstinence period and pregnancy rates after IUI.

Several studies suggested performing IUI with sperm samples obtained in a shorter abstinence period than recommended by WHO. However, there isn't enough research on this issue in the literature. Moreover, there is no specific prospective clinical research examining the relationship of ejaculatory abstinence period and sperm DNA fragmentation in IUI cycles. The aim of this study was to report the effect of ejaculatory abstinence on sperm DNA fragmentation and pregnancy rates in IUI cycles, as well as the correlation between the two

ELIGIBILITY:
Inclusion Criteria:

* Infertility for more than 12 months
* Diagnosed as unexplained infertility
* Female age between 20 and 40 years
* Regular menstrual cycles
* Mid-luteal progesterone levels of >3 ng/ml
* Basal FSH <12 mIU/ml, AMH >1ng/ml
* Body mass index (BMI) 19-35 kg/m2
* No pelvic pathology documented by transvaginal ultrasound and bilateral tubal patency diagnosed by hysterosalpingography
* Normal semen parameters according to WHO criteria

Exclusion Criteria:

* Any endocrine and pelvic pathology
* PCOS (polycystic ovarian syndrome)
* Known endometriosis history
* Prior pelvic surgery
* Persistent ovarian cysts.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Couples with the diagnosis of unexplained infertility.
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | The pregnancy test was done 14 days after intrauterine insemination. If the test was positive, transvaginal ultrasonography was performed at 6-7 weeks of gestation.
  The presence of one or more gestational sacs on transvaginal ultrasonography was described as clinical pregnancy.

SECONDARY OUTCOMES:
Sperm DNA fragmentation percentage | On the day of IUI, semen samples were obtained and the sperm DNA fragmentation was measured by the TUNEL method in the inseminated sperm.
  Sperm DNA fragmentation rate assessed by TUNEL assay.

CONTACTS AND LOCATIONS:
Overall Officials: CIHAN KABUKCU, M.D., Principal Investigator — Department of Obstetrics and Gynecology - Infertility Center
Locations (1):
- Pamukkale University Faculty of Medicine, Obstetrics and Gynecology Department, Infertility Center, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jurema MW, Vieira AD, Bankowski B, Petrella C, Zhao Y, Wallach E, Zacur H. Effect of ejaculatory abstinence period on the pregnancy rate after intrauterine insemination. Fertil Steril. 2005 Sep;84(3):678-81. doi: 10.1016/j.fertnstert.2005.03.044. PMID 16169402
- [Background] Marshburn PB, Alanis M, Matthews ML, Usadi R, Papadakis MH, Kullstam S, Hurst BS. A short period of ejaculatory abstinence before intrauterine insemination is associated with higher pregnancy rates. Fertil Steril. 2010 Jan;93(1):286-8. doi: 10.1016/j.fertnstert.2009.07.972. Epub 2009 Sep 3. PMID 19732887
- [Background] Thomson LK, Zieschang JA, Clark AM. Oxidative deoxyribonucleic acid damage in sperm has a negative impact on clinical pregnancy rate in intrauterine insemination but not intracytoplasmic sperm injection cycles. Fertil Steril. 2011 Oct;96(4):843-7. doi: 10.1016/j.fertnstert.2011.07.356. Epub 2011 Aug 11. PMID 21839433
- [Derived] Kabukcu C, Cil N, Cabus U, Alatas E. Effect of ejaculatory abstinence period on sperm DNA fragmentation and pregnancy outcome of intrauterine insemination cycles: A prospective randomized study. Arch Gynecol Obstet. 2021 Jan;303(1):269-278. doi: 10.1007/s00404-020-05783-0. Epub 2020 Sep 9. PMID 32902676